CLINICAL TRIAL: NCT04020380
Title: A Single Arm, Open-label Exploratory Clinical Trial of Azithromycin in Pulmonary Sarcoidosis
Brief Title: Azithromycin a Treatment for Pulmonary Sarcoidosis
Acronym: CAPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC2019
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Sarcoidosis, Pulmonary
MeSH Terms: conditions — Sarcoidosis, Pulmonary | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: single centre, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azithromycin 250 mg (Experimental): Azithromycin, 250 mg capsules once a day for a total of 3 months
  Interventions: Drug: Azithromycin 250Mg Capsule

INTERVENTIONS:
Drug: Azithromycin 250Mg Capsule — 250 mg OD

SUMMARY:
Patients with sarcoidosis need treatment options that effectively control their disease without causing undesirable side effects. An appealing strategy is to repurpose existing drugs which possess beneficial immune modulating activity and are safe for long-term use. Recently, increased activity of the mTOR intracellular signalling pathway in inflammatory cells has emerged as a key driver of granulomatous inflammation in mouse models and patients with sarcoidosis. The macrolide antibiotic azithromycin directly inhibits mTOR activity in inflammatory cells, making it a prime target for drug repurposing in sarcoidosis. Azithromycin has an acceptable tolerability profile when used for long-term treatment of other chronic respiratory disease Single centre open label clinical trial of oral azithromycin 250 mg once daily for 3 months in 20-30 patients with pulmonary sarcoidosis.

The Investigator have opted for an open label study because this will be the first study of azithromycin in sarcoidosis. Trial assessments will be performed according to standards of Good Clinical Practice with assessments at baseline, 1, and 3 months. All other clinical care, investigations, and treatment (if indicated) will remain the responsibility of the treating physician and based on clinical MDT consensus decisions.

DETAILED DESCRIPTION:
Disease behavior in sarcoidosis is variable and difficult to predict. Spontaneous improvement may occur, but even then evidence of persistent low grade granulomatous inflammation is common and disabling symptoms such as fatigue may persist. Patients with milder chronic sarcoidosis may suffer significant symptoms and disability, but active monitoring and supportive care are the only currently suitable management options. Recurrence after remission is a problem, with some patients suffering from chronic ill health, progressive disease and fibrosis, potentially leading to organ failure and death or transplantation. Management is further complicated because some patients with symptomatic, progressive sarcoidosis have a high burden of granulomatous disease, often affecting the lungs, whereas other patients have limited disease in a dangerous location such as the heart or nervous system.

Cure is not a realistic option whilst the cause(s) of sarcoidosis remain unknown. Ideally, treatment should be aimed at preventing or slowing progression to irreversible fibrosis and organ failure, reducing symptoms, and improving quality of life. The evidence that currently used treatments achieve these aims is weak, and the risk of adverse effects is concerning for patients and may outweigh perceived benefits. Treatment with corticosteroids is suppressive rather than curative, and guidelines recommend at least 1 years' therapy for patients with progressive disease. In the BTS sarcoidosis study, long term corticosteroids given to patients with non-resolving pulmonary disease after six months' initial observation improved lung function and chest x-ray appearances by a small amount. Importantly, of patients who were given early steroids for troublesome symptoms, almost half were still taking steroids 5 years later. Yet whether steroids prevent fibrosis or improve clinically meaningful outcomes that are important to patients in the longer term is unknown. Worryingly, there is evidence that early steroid therapy may promote more aggressive disease later on. Side effects of steroid therapy are often distressing and disfiguring, and sometimes serious or fatal. When sarcoidosis is refractory to steroid treatment, second line immunomodulators such as methotrexate, azathioprine, or mycophenolate are commonly prescribed based on their efficacy in treating rheumatic diseases, and are recommended in guidelines. In sarcoidosis, the best evidence is that they are steroid sparing (i.e. permit a lower dose of corticosteroid to be used). As with steroids, long term benefits have not been demonstrated and liver and bone marrow toxicity is a concern, requiring regular blood testing.

Whilst a unifying cause of sarcoidosis remains elusive, it has been established that inflammatory cells including T lymphocytes, monocytes, and macrophages become hyper-activated in the lungs and peripheral blood. Recently, using mouse models it has been shown that chronic signalling through the mTOR complex 1 (mTORC1) in macrophages pathway drives the formation of sarcoid-like granulomas that closely mimic non-resolving sarcoidosis in humans. mTOR (mammalian/mechanistic target of rapamycin) links growth factors and availability of amino acids to protein synthesis and cell growth, proliferation, and differentiation. mTOR activity and gene targets correlating to sarcoidosis progression in lung biopsies have implicated a potential role for targeting mTOR in human disease. These datasets indicate a key role for mTOR pathways and the metabolic status of tissue macrophages in triggering and driving disease pathology.

The macrolide antibiotic azithromycin is immunomodulatory and anti-bacterial, both of which are plausible beneficial properties in sarcoidosis. Many studies have implicated bacteria as triggers for sarcoidosis, and although convincing evidence implicating a specific organism is lacking, improvements in sarcoidosis have been described in antibiotic combination studies that included azithromycin. Beneficial immunomodulatory properties of macrolides became apparent in the treatment of Asian diffuse panbronchiolitis, where reduced inflammatory cytokine production in several cell types was demonstrated. Recently, it has been determined that azithromycin directly suppresses mTOR activity in a subset of T lymphocytes (CD4+ T-cells).

Patients with pulmonary sarcoidosis need treatment options that effectively modulate disease activity, reduce risk of disease progression, and improve symptoms and quality of life, with an acceptable side effect profile. Azithromycin is a cheap, readily available generic drug. Long term treatment with azithromycin has been shown to be safe in other chronic lung diseases. Azithromycin is preferable to other macrolide antibiotics because of its safety data for long term use, once daily administration, and lack of inhibition of liver CYP3A isoenzymes. The safety profile of azithromycin makes it preferable to non-antibiotic macrolide mTOR inhibitors such as rapamycin (sirolimus, used to treat transplant rejection)) and everolimus (an anti-cancer drug). Whether azithromycin will benefit patients with sarcoidosis can only be answered definitively by a large multicenter clinical trial. The Investigators proposed exploratory study aims to facilitate this aim by exploring mechanisms and evaluating potential blood biomarkers, and assessing feasibility of a subsequent large clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* • Males or females, of any race, between 18 and 80 years of age, inclusive;

  * Able to speak, read, and understand English;
  * Able to provide written informed consent;
  * Able to communicate effectively with the Investigator and other study centre personnel and agree to comply with the study procedures and restrictions.
  * Clinician diagnosis of pulmonary sarcoidosis;
  * If a female of child-bearing potential (i.e., have not undergone a hysterectomy or bilateral oophorectomy) or not post-menopausal (defined as no menses for at least 12 months), agree to use acceptable birth control (defined in Section 6.3) from screening through to the follow up visit;

Exclusion Criteria:

* • Hypersensitivity to azithromycin or another macrolide antibiotic (e.g. erythromycin, clarithromycin) or excipients (see 7.4)

  * History of signficant cardiac arrhythmia
  * Personal or family history of congenital long QT syndrome;
  * Prolonged QTc interval on 12-lead ECG
  * Signficant liver disease
  * Evidence of acute bacterial infection
  * Clinically significant bronchiectasis
  * Requiring concomitant therapy with prohibited medications (see Section 7.5)
  * Pregnant or breastfeeding;
  * Treatment with an investigational drug or biologic within 30 days preceding the first dose of study medication or plans to take another investigational drug or biologic within 30 days of study completion;
  * Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the Investigator or Sponsor, would make the subject inappropriate for entry into this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
change in 24 hr cough counts from baseline | 3 months
  24n hr cough monitoring with ambulatory cough monitor will be performed at baseline and at 1mth and 3 months post treatment

SECONDARY OUTCOMES:
Mean Change in severity of cough from baseline | 3 months
  Severity of cough will be scored on a visual anolgue scale at baseline and at 1month and 3 months post treatment
Mean Change in urge to cough from baseline | 3 months
  Urge to cough will be scored on a visual analogue scale at baseline and at 1 month and 3 months post treatment
Mean Change in Leicester cough questionnaire total score from baseline | 3 months
  The Leicester cough questionnaire will be performed at baseline and at 1 month and 3 months post treatment.
Mean Change in Kings sarcoidosis questionnaire total score from baseline | 3 months
  Kings sarcoidosis questionniare will be completed at baseline and compared with that at 1 month and 3 months post azithromycin

CONTACTS AND LOCATIONS:
Overall Officials: Simon Hart, MD, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Respiratory Medicine Clinical trials Unit, Cottingham, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No